CLINICAL TRIAL: NCT02663882
Title: Self-Control and Adult Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Responsible Party: Principal Investigator, Andrea Weinberger, Associate Professor, Yeshiva University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-5479
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Smoking
Keywords: smoking; self control
MeSH Terms: conditions — Smoking; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- smoking-related self control task (Experimental): self control practice - smoking related task
  Interventions: Behavioral: self control practice - smoking related task
- Non-smoking-related self control task (Active Comparator): self control practice - non-smoking related task
  Interventions: Behavioral: self control practice - non-smoking related task

INTERVENTIONS:
Behavioral: self control practice - smoking related task — participants will be asked to practice a smoking-related self control task for 7 days: they will be asked to resist smoking when they have cravings as much as possible during the day
  Arms: smoking-related self control task
Behavioral: self control practice - non-smoking related task — participants will be asked to practice a non-smoking-related self control task for 7 days: they will be asked to keep a straight posture as much as possible during the day
  Arms: Non-smoking-related self control task

SUMMARY:
The purpose of this study is to learn more about self-control and adults who smoke cigarettes. It has been suggested that people can improve self-control by practicing tasks that require the use of self-control (such as delaying cigarettes or sitting up as straight as possible). The goal of this study is to learn about whether scores on self-control and other measures will change after one week of practicing self-control tasks at home. We believe that adults who smoke cigarettes will show better self-control after practicing tasks for a week.

DETAILED DESCRIPTION:
The purpose of this pilot study is to examine a smoking-related self-control task and smoking behavior in adult smokers who are not motivated to quit smoking.

This pilot study will have a between-subjects design. All participants will be asked to complete two study appointments. First, they will complete a baseline appointment where they will review consent procedures. Participants who complete the consent forms will then be asked to fill out measures of demographics, smoking, and self-control. Smoking will be confirmed using expired breath carbon monoxide (CO) levels taken using a CO monitor. At that appointment participants will be randomly assigned to complete one of two self-control tasks: a task that is related to smoking (e.g., giving instructions to delay smoking when they have a craving) or a task that is not related to smoking (e.g., participants will be instructed to try to maintain the best posture possible (e.g., sit up straight, walk with good posture) as much as possible throughout each day Random assignment will be done using a random number generator and 50% of participants will be assigned to the smoking task while the other 50% will be assigned to the non-smoking task. Study staff will received standardized instructions to read to each participant about the task that they are assigned to practice during the week. Participants will be asked to practice their assigned self-control task every day for a week and to complete a brief series of questions about the effort and time spent practicing the task that day along with the number of cigarettes they smoked that day. After one week, participants will return for the second study appointment where they will report on their effort and time spent practicing the self-control tasks and complete additional measures of smoking and self-control.

ELIGIBILITY:
Inclusion Criteria:

1. Be adults who are 18 years of age or older
2. Currently smoke ≥10 cigarettes per day biochemically confirmed by an expired breath carbon monoxide (CO) level ≥8
3. Report that they are not currently attempting to quit smoking and not currently receiving smoking cessation treatment (e.g., counseling, nicotine replacement therapy, bupropion, varenicline)
4. Have the capacity to give informed consent
5. Be English-speaking.

Exclusion Criteria:

1. Children under the age of 18
2. Non-English speakers
3. Those who do not have the capacity to consent will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea H Weinberger, PhD, Principal Investigator — Yeshiva University
Locations (1):
- Smoking and Nicotine Dependence Research Laboratory, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task
Started | 39 | 36
Completed | 35 | 34
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.1) | 46.8 (11.3) | 44.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 28 | 28 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 27 | 29 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 22 | 48
  White | 8 | 8 | 16
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 36 | 75

OUTCOME MEASURES:

1. Primary Outcome: Self- Control as Measured by the Change in the Length of Time Participants Can Hold a Hand-grip at Baseline and Follow-up (One Week After Baseline)
Description: Participants were instructed to squeeze a hand-grip exerciser as long as possible and research staff used a stopwatch to time the length of time that the hand-grip is squeezed. A wad of paper was inserted between the handles of the hand-grip and timing stopped when the paper fell from the hand-grip indicating that the participant had released the hand-grip. The hand-grip was held before and after a thought suppression exercise that was meant to diminish self-control in order to control for individual hand strength.
  Self-control was measured as the difference in the length of time holding the hand-grip before and after the thought suppression exercise at each appointment (baseline and one week followup).
  Change in self-control due to task practice was measured as [self-control at the second study appointment one week after the first appointment] minus [self-control at the first study appointment].
Time Frame: Baseline, one week followup after baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task
Number analyzed (Participants) | 35 | 34
seconds
  data from baseline appointment | -9.36 (103.42) | 2.76 (80.82)
  data from second appointment, one week after baseline | -4.32 (109.14) | 42.88 (179.95)
Statistical Analysis 1: Comparison: Smoking-related Self Control Task vs Non-smoking-related Self Control Task; The non-smoking-related self control task was the comparison group in relation to the smoking-related self control task; Test type: Superiority; p = 0.503, ANOVA — the a priori threshold for statistical significance was p<0.05

2. Secondary Outcome: Self-Control as Measured by the Change in Self-reported Overall Self-Control at Baseline and Follow-up
Description: Self-control was measured using the investigator-developed Overall Self Control question (1 item):
  Participants were asked: How would you rate your overall level of self-control on a scale from 0 (I have no self-control) to 10 (I have complete self-control)?
  The response scale was a 10-point Likert scale ranging from 0 (I have no self-control) to 10 (I have complete self control).
  Higher scores indicated higher self control.
Time Frame: 2 assessments of this item over one week (baseline appointment, follow up appointment 1 week after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task
Number analyzed (Participants) | 35 | 34
score on a scale
  baseline | 6.1 (2.4) | 6.3 (4.5)
  followup | 6.5 (2.1) | 6.9 (5.2)
Statistical Analysis 1: Comparison: Non-smoking-related Self Control Task; The non-smoking-related self control task was the comparison group in relation to the smoking-related self control task; Test type: Superiority; p = 0.765, ANOVA — the a priori threshold for statistical significance was p<0.05

3. Secondary Outcome: Change in Smoking Quantity (Cigarettes Smoked Per Day) Measured at Baseline and at Follow-up
Description: Change in self-reported average number of cigarettes smoked per day from study appointment 1 (baseline) to study appointment 2 (one week later).
  There is no official title to this item (cigarettes per day). Participants were asked to respond to this investigator-written question: "How many cigarettes each day do you smoke right now?"
  The response scale was open ("I smoke ________ cigarettes each day that I smoke") so that participants could write in any number of cigarettes. At baseline, there was no official minimum value but participants had to report smoking 10 cigarettes a day as part of the inclusion criteria for the study. There was no maximum response option provided. For the followup assessment (one week after baseline), participants were asked the same questions and there was no minimum or maximum response options provided.
  Higher numbers indicate a greater number of cigarettes smoked each day
Time Frame: Baseline, follow up appointment one week after baseline
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task
Number analyzed (Participants) | 35 | 34
cigarettes per day
  baseline | 13.1 (4.1) | 12.0 (5.7)
  followup appointment one week after baseline | 12.0 (5.7) | 13.2 (4.3)
Statistical Analysis 1: Comparison: Smoking-related Self Control Task vs Non-smoking-related Self Control Task; The non-smoking-related self control task was the comparison group in relation to the smoking-related self control task; Test type: Superiority; p = 0.717, ANOVA — the a priori threshold for statistical significance was p=0.05

4. Secondary Outcome: Change in Expired Breath Carbon Monoxide Level
Description: Change in a biochemical measure of smoking (expired breath carbon monoxide level) from study appointment 1 (baseline) to study appointment 2 (one week later)
  This measure is not a scale. Participants provide a breath sample into a carbon monoxide monitor and the monitor provides a number from 0 and up in ppm (parts per million). Higher numbers indicate greater levels of carbon monoxide and this level is used as a proxy for amount of recent smoking (higher numbers indicating greater recent smoking).
Time Frame: Baseline, follow up one week after baseline
Measure: Mean (Standard Deviation); unit: ppm (parts per million)
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task
Number analyzed (Participants) | 35 | 34
ppm (parts per million)
  baseline | 18.4 (6.4) | 16.6 (6.6)
  followup (one week after baseline) | 16.8 (10.4) | 16.8 (5.5)
Statistical Analysis 1: Comparison: Smoking-related Self Control Task vs Non-smoking-related Self Control Task; The non-smoking-related self control task was the comparison group in relation to the smoking-related self control task; Test type: Superiority; p = 0.302, ANOVA — the a priori threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: 1 week (baseline appointment and appointment one week after baseline)
Description: does not differ
Arm/Group | Smoking-related Self Control Task | Non-smoking-related Self Control Task
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 0/39 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02663882/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT02663882/Prot_SAP_001.pdf